CLINICAL TRIAL: NCT03172117
Title: Follow-up Study of Safety and Efficacy in Subjects Who Completed NEUROSTEM® Phase-I/IIa Clinical Trial.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-CR-010-F/U
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NEUROSTEM® (hUCB-MSCs)- low dose (Experimental): human umbilical cord blood derived mesenchymal stem cells Low dose: 1 x 10^7cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  Interventions: Biological: human umbilical cord blood derived mesenchymal stem cells
- NEUROSTEM® (hUCB-MSCs) - high dose (Experimental): human umbilical cord blood derived mesenchymal stem cells High dose: 3 x 10^7 cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  Interventions: Biological: human umbilical cord blood derived mesenchymal stem cells
- Placebo (Placebo Comparator): normal saline 2mL, doses separated by 4 weeks for a total of 3 doses
  Interventions: Other: Normal saline 2mL

INTERVENTIONS:
Biological: human umbilical cord blood derived mesenchymal stem cells — Low dose: 1 x 10^7cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  High dose: 3 x 10^7cells/2mL 3 repeated intraventricular administrations via an Ommaya Reservoir at 4 week intervals
  Other Names: NEUROSTEM®
  Arms: NEUROSTEM® (hUCB-MSCs) - high dose; NEUROSTEM® (hUCB-MSCs)- low dose
Other: Normal saline 2mL — Normal Saline at 4 week intervals via an Ommaya Reservoir, for a total of 3 administrations
  Arms: Placebo

SUMMARY:
A long-term follow-up study to obtain safety and efficacy data in subjects who completed phase 1/2a clinical trial of NEUROSTEM® (NCT02054208), comparing NEUROSTEM and placebo groups for up to 36 months after the initial administration in patients suffering from Alzheimer's disease

DETAILED DESCRIPTION:
The subjects will be followed up at 12-month, 24-month, and 36-month (phone call) after the initial administration of NEUROSTEM®.

ELIGIBILITY:
Inclusion Criteria:

* Assessment of safety and exploratory treatment efficacy in subjects who were enrolled and completed phase 1/2a clinical trial of NEUROSTEM®.
* Subjects who have been treated with either NEUROSTEM® or placebo at least 12 months ago.
* Subjects who voluntarily decided to participate and signed the consent form after receiving explanations on the clinical trial (in case it is difficult for the participant to sign, the consent of the legal representative)

Exclusion Criteria:

* Subjects who were not enrolled in phase 1/2a clinical trial of Neurostem® for assessing safety and exploratory treatment efficacy
* Other subjects, excluding those listed above, who were deemed unsuitable by the PI

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Change from the baseline in ADAS-Cog | 24 month after the first dose
  Alzheimer's Disease assessment Scale-Cognitive Subscale

SECONDARY OUTCOMES:
Change from the baseline in S-IADL | 24 month after the first dose
  Seoul Instrumental Activities of Daily Living
Change from the baseline in K-MMSE | 24 month after the first dose
  Mini Mental State Exmination Korean version
Change from the baseline in CGA-NPI | 24 month after the first dose
  Caregiver-administered Neuropsychiatric Inventory
ADAS-Cog Response Rate | 24 month after the first dose
  the ADAS-cog score at 24 month after the first administration compared to the baseline
Change in CDR-SOB | 24 month after the first dose
  Clinical Dementia Rating-Sum of Box
Change in CIBIC-plus | 24 month after the first dose
  The Clinician's Interview Based Impression of Change-plus
Change in Florbetaben-PET | 24 month after the first dose
  Florbetaben - Pittsburgh Compound B-positron emission tomography
Change in FDG-PET (CMRglc: regional cerebral metabolic rate for glucose) | 24 month after the first dose
  fluorodeoxyglucose positron emission tomography
Change from baseline in MRI (DTI mapping) | 24 month after the first dose
  MRI Analysis
Change from the baseline in CSF biomarkers | 24 month after the first dose
  biomakrer analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee NK, Jang H, Choi Y, Hwangbo S, Lee S, Lee JI, Kim YJ, Chin J, Chang JW, Seo SW, Son HJ, Choi SJ, Na DL, Kim HJ. Mesenchymal Stem Cells With Adjuvant Dexamethasone in Patients With Alzheimer's Disease: A Phase IIa Trial. Dement Neurocogn Disord. 2025 Oct;24(4):272-285. doi: 10.12779/dnd.2025.24.4.272. Epub 2025 Oct 24. PMID 41220869
- [Derived] Kim HJ, Cho KR, Jang H, Lee NK, Jung YH, Kim JP, Lee JI, Chang JW, Park S, Kim ST, Moon SW, Seo SW, Choi SJ, Na DL. Intracerebroventricular injection of human umbilical cord blood mesenchymal stem cells in patients with Alzheimer's disease dementia: a phase I clinical trial. Alzheimers Res Ther. 2021 Sep 14;13(1):154. doi: 10.1186/s13195-021-00897-2. PMID 34521461